CLINICAL TRIAL: NCT06872827
Title: Effect of Herbal Toothpaste Versus Conventional One on Black Stains in a Group of Egyptian Children: A Randomized Controlled Study
Brief Title: Effect of Herbal Toothpaste Versus Conventional One on Black Stains
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Mohamed Farouk Rashed, Researcher of Pediatric Dentistry, Orthodontics and Pediatric Dentistry Department, Oral and Dental Research Institute National Research Centre, National Research Centre, Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 341
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Black Stains
Keywords: black stains; bacteria; herbal; child

STUDY DESIGN:
Intervention Model Description: Randomized controlled parallel triple blinded study
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple (Participant, Investigator, Outcomes Assessor) Blinding to the child participants and legal guardian of each participating child, inter examiner and statistician. The operator and the child were blinded to the intervention from the beginning till teeth polishing. Blinding cannot be done during application of toothpaste because of clear visual differences between these toothpastes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Herbal toothpaste
  Interventions: Drug: Herbal toothpaste
- Control (Active Comparator): Signal toothpaste
  Interventions: Drug: Herbal toothpaste

INTERVENTIONS:
Drug: Herbal toothpaste — Intervention
  Other Names: Dabur Red toothpaste

SUMMARY:
Twenty eight children with black stains on their teeth were divided into 2 groups of toothpaste to assess their effect on parental satisfaction, recurrence rate of black stains and change in number of bacteria before and after treatment

DETAILED DESCRIPTION:
TChildren will be enrolled in the study from the outpatient dental Clinic, Medical Centre of Excellence, National Research Centre, Egypt. After professional polishing of blacks stains subjects will be randomly assigned in two groups of equal number (n=28; subdivided to 14 in each group).

The test group will use herbal toothpaste (Dabur Red); (Garik powder (Red ochre), Pippali (Piper longum), Maricha (Piper nigrum), Sunthi (Zingiberofficinale), Tomarbeej (Zanthoxylumarmatum), Karpoor (Cinnamomumcamphora), Laungka Tail (Oil of Syzygiumaromaticum) and Pudinasatva (Menthapiperita).); the control group will use toothpaste with sodiumfluoride toothpaste (Signal). (Aqua, Hydrogenated Starch Hydrolysate, Hydrated Silica, PEG-32, Zinc Citrate, Sodium Lauryl Sulfate, Aroma, MenthaPiperita Oil, Rosmarinus Officinalis Leaf Oil, Cellulose Gum, Sodium Fluoride, Sodium Saccharin, Glycerin, Sodium Bicarbonate, Limonene, CI 74260).

Both test and control groups will use the assigned toothpaste twice a day for 2 months. The study will be double-blinded; sequentially numbered, opaque, sealed envelopes containing the test or the control tooth paste will be prepared.

At the beginning of the study, all subjects will complete a questionnaire including questions regarding socio-demographic variables such as age and sex. Subjects with BS(test and control groups) will also asked about oral hygiene habits such as type of dental brush (manual or electric), dietary habits such as iron supplementation and type of drinking water consumed (tap or mineral water).

The test and control subjects will receive training for home dental hygiene at enrollment and will be contacted by phone every 2 weeks for 2 months to ensure adherence to the protocol and record any recurrence of black stains.

All enrolled subjects will be followed at the Dental Clinic, National Research Centre, Egypt. The study will be consistent with good clinical practices in accordance with the Ethical Principles of the "64th World Medical Association Declaration of Helsinki". All Participants parents will sign a written informed consent before joining the study after brief explanation of all procedures and time table. A verbal assent will be taken from the child before intervention.

Clinical Examination and Samples Collection:

All subjects with BS (both test and control group) will have intraoral examination and professional oral prophylaxis at the enrollment by the same operator. Intraoral photographs will be collected. Clinical evaluation of BS will be assessed carefully to exclude other causes of dental stains. Mean number of Decayed, Missing, and Filled primary and permanent Teeth index (DMFT/deft) will be also calculated.

Salivary Samples collection Five ml of unstimulated saliva samples from all participants from both test and control groups will be collected in a sterile 15 ml falcon tube according to standard procedures. Samples will be collected before using the herbal and conventional toothpaste and after 2 months of their regular use.

DNA extraction Total DNA from the saliva samples of all participants will be done using genomic commercial DNA extraction kit, according to the supplier's instructions. The integrity of DNA will be checked using agarose gel electrophoresis and the concentration and the purity of DNA samples will be checked using NanoDrop spectrophotometer.

Quantification of bacterial species using qRT-PCR Two species of cariogenic bacteria; Streptococcus mutans and Lactobacillus casei are selected to be involved in this study. In addition, two species of chromogenic bacteria; Actinomyces naeslundii and Prevotella melaninogenica will be included in the present study. The sequences of primers of the selected bacterial species; F=TCGCGAAAAAGATAAACAAACA and R=GCCCCTTCACAGTTGGTTAG for (Streptococcus mutans), F=TTAAAGCCATTCTCAGTTCGGA and R=TACGGCTACCTTGTTACGACTT for (Lactobacillus casei) (12). An-F3: CTGCTGCTGACATCGCCGCTCGTA and An-R3: TCCGCTCGCGCCACCTCTCGTTA for (Actinomyces naeslundii), Pm-F3: TGACCGTAAGAAGAAGTTGCCTGTA and Pm-R3: TTGCGACCGATAGCTGCCTTCATA for (Prevotella melaninogenica) (13). Quantification of the selected bacterial species will be carried out using SYBR green master mix, specific primers, DNA and complete the volume of the reaction mixture using sterile RNase and DNase free water. The reaction will be done using real-time polymerase chain reaction in RT-PCR device.

ELIGIBILITY:
Inclusion criteria:

1. Children 6 to 12 years
2. Free medical history.
3. Presence of black stains covering at least two teeth.
4. Good oral hygiene.

Exclusion criteria:

1. Children on iron supplements
2. Presence of intrinsic stains or fluorosis
3. Children using electric toothbrush.
4. Children took mouthwash or antibiotic in the last month.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Parental satisfaction using Likert scale regarding both interventions of management of black stains (Each response was scored as follows: (5) strongly agree, (4) agree, (3) neutral, (2) disagree and (1) strongly disagree). | After 2 months
  using Likert scale regarding both interventions of management of black stains (Each response was scored as follows: (5) strongly agree, (4) agree, (3) neutral, (2) disagree and (1) strongly disagree).

SECONDARY OUTCOMES:
Recurrence of black stains | After 2 months
  Recurrence rate of black stains

OTHER OUTCOMES:
Change in number of bacteria before and after treatment | After 2 months
  Change in number of bacteria before and after treatment using qRT-PCR regarding both interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed F Rashed, Researcher, Study Director — National Research Centre, Egypt
Locations (1):
- National Research Centre, Dokki, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No